CLINICAL TRIAL: NCT03655639
Title: Evaluating Cardiorespiratory Development in Premature Babies
Brief Title: Local Version of the Multi-center PREVENT Study Evaluating Cardio-respiratory Instability in Premature Infants
Status: Active, not recruiting | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Northwestern Memorial Hospital (Other); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-1178; U01HL133704 (NIH)
Record Dates: First submitted 2018-08-22; First posted 2018-08-31 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal DNA swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature Birth: Premature babies born under 29 weeks gestational age, admitted into the neonatal intensive care unit within 7 days of life.

SUMMARY:
Infants who are born prematurely have immature nervous and cardiorespiratory systems. These are systems infants use to breathe, to move oxygen throughout their bodies, and to maintain safe and stable levels of oxygen and carbon dioxide. The goal of this study is to better understand how these immature systems affect long term development, such as brain, heart, and motor function (movement) with several innovative, integrated physiological measures. We hope this will allow us to begin to find better ways to help premature infants breathe and to optimize their development.

DETAILED DESCRIPTION:
The broad long-term objective is to use comprehensive state-of-the-art, high-fidelity monitoring to investigate physiological biomarkers of autonomic neurorespiratory maturation with integrated analysis of autonomic nervous system (ANS) responses in preterm infants, and to evaluate their role in ventilatory instability, bronchopulmonary dysplasia (BPD), and co-morbidities including neurodevelopment in the 1st year of life. SPECIFIC AIM 1 will establish the spectrum and developmental trajectory of ANS maturation/function using high-resolution physiologic recordings of ventilatory, cardiovascular, and cerebrovascular measures during typical daily activity (28, 32 and 36 weeks (wks) post-menstrual age (PMA)(up to 24-hour recordings) and at 3 and 12 months (mos) corrected age (CA)(4-hour recordings). Aim 1 tests the hypothesis that individual and integrated metrics of ANS function will demonstrate maturational patterns that impart resilience or vulnerability to environmental challenges. SPECIFIC AIM 2 will determine respiratory and neurodevelopmental morbidity throughout the 1st year of life using clinically applicable outcome measures and associate morbidity with ANS development and function using a Respiratory Morbidity Severity Score (RMSS), need for respiratory support, medications, or hospitalization, Bayley Scales of Infant Development III (6, 12 mos), Neurological, Sensory, Motor, Developmental Assessment (NSMDA)(3, 6, 12 mos), and early measures of evoked-auditory potentials (EAP)(28, 32, 36 wks PMA; 3, 12 mos CA) and General Movement Assessments (GMA)(28, 32, 36 wks; 3 mos). Aim 2 tests the hypothesis that infants demonstrating delayed ANS maturation or vulnerability to endogenous challenges will require more respiratory interventions and will demonstrate developmental delays in the 1st year of life. SPECIFIC AIM 3 will determine endotypes of autonomic neurorespiratory stability and maturation through trajectory analysis and integrated physiological modeling. Aim 3 tests the hypothesis that trajectory analysis will reveal 3 autonomic maturation patterns [1) "normal" maturation with ability to withstand environmental perturbations; 2) "normal" maturation without ability to withstand environmental perturbations; and 3) delayed or disordered maturation with inability to maintain physiologic stability in absence of environmental perturbations] that will be associated with severity of respiratory morbidity and neuromotor impairment at 1 year. This novel approach will establish the role of autonomic neurorespiratory maturation in stability of oxygenation throughout the 1st year of life, provide insight into BPD pathogenesis, allow prospective identification of at-risk infants, and permit development of mechanism-specific interventions with potential to impact thousands of families and billions in healthcare cost/year in the U.S., alone.

In addition to lung-independent mechanisms of respiratory dysfunction, this study aims to investigate lung-independent mechanisms of pulmonary hypertension (PH). Typically thought to be a secondary effect of primary lung structural development and/or hypoxia, up to 40% of infants with chronic respiratory dysfunction develop pulmonary hypertension (PH) and increased risk for mortality. However, we and others found that 10-30% of premature infants who develop PH did not have clinical evidence of respiratory dysfunction, suggesting pulmonary vascular mechanisms that are independent of clinically apparent respiratory disease. Multiple molecular mechanisms are postulated by which hypoxia results in PH, but preliminary data from our group and others suggest a role for Fibroblast Growth Factor 2 (FGF2) and FGF receptors 1 and 2 (FGFR1, FGFR2) signaling in the development of pulmonary vascular remodeling in PH. Thus, by serially using sensitive echocardiographic measures of Right Ventricular-Pulmonary Arterial (RV-PA) coupling, we can quantify hypoxic exposure and RV-PA axis dysfunction and we will couple these clinical measurements of FGF2 signaling. We hypothesize that recurrent hypoxic exposure of dysmature pulmonary vasculature in premature newborns results in RV-PA axis dysfunction and pulmonary hypertension that is mediated by FGF2 signaling and is independent of clinically apparent lung disease.

ELIGIBILITY:
Inclusion Criteria:

* birth between 24 and 29 weeks of gestation
* less than 1 week of age

Exclusion Criteria:

* known congenital anomalies
* imminent death
* factors that preclude reliable follow-up

Ages: 24 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature babies born under 29 weeks of gestational age, who are admitted into the neonatal intensive care unit within a week of birth.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory coupling between 28 weeks postmenstrual age and 1 year | 1 year
  Average cross-spectral coherence between heart rate and respiratory rate summed within the high frequency band (above 0.15 Hz; ratiometric units). Higher coherence indicates better coupling.

SECONDARY OUTCOMES:
Neurodevelopmental outcomes as measured with the Neurological, Sensory, Motor, Developmental Assessment (NSMDA) functional grade | 1 year
  6 subtests are scored individually (1-5 with 1 being normal, 5 with profound disability) and added together - normal 6-8, 9-11 minimal dysfunction, 12-14 mild problems, 16-19 moderate disability, 20-24 severe disability and 25-30 multiple, severe or profound disabilities.

OTHER OUTCOMES:
Change in right ventricle-pulmonary circulation (RV-PC) axis function between 32 and 36 weeks postmenstrual age | 36 weeks postmenstrual age
  echocardiographic measurements of pulmonary artery acceleration time (PAAT, milliseconds), where values less than 43 msec are indicative of RV-PC axis dysfunction
Changes in circulating levels of fibroblast growth factor 2 (FGF2) and granulocyte macrophage colony stimulating factor (G-CSF) between 32 and 36 weeks postmenstrual age | 36 weeks postmenstrual age
  comparison of FGF2 and G-CSF levels as measured by immunoassay between infants with and without RV-PC axis dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Hamvas, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois